CLINICAL TRIAL: NCT05646303
Title: A 24-Week, Multicentre, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Clinical Trial to Evaluate Efficacy and Safety of Psilocybin-Assisted Psychotherapy in Adults With Alcohol Use Disorder (AUD)
Brief Title: Psilocybin-Assisted Psychotherapy in Adults With Alcohol Use Disorder (AUD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clairvoyant Therapeutics (Industry)
Collaborators: Optimapharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLA PSY 201
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): 2 oral doses of 25mg psilocybin capsules
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator): 2 oral doses of placebo (microcrystalline cellulose) capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — Psilocybin and psychotherapy
  Arms: Psilocybin
Drug: Placebo — Placebo and psychotherapy
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate treatment with psilocybin and psychotherapy for the treatment of people with Alcohol Use Disorder (AUD). The main question[s] it aims to answer are:

* Does treatment with psilocybin and therapy help reduce alcohol consumption more than placebo and therapy?
* Is treatment with psilocybin and therapy safe for participants?

Participants will

* Attend 13 study visits
* Take part in therapy sessions including 2 treatment sessions with either psilocybin or placebo
* Record their daily alcohol consumption on study specific device

Researchers will compare psilocybin and placebo groups to see if alcohol consumption is decreased.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe diagnosis of AUD as measured by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria using Structured Clinical Interview for DSM-5 by the investigator.
* Expressed a wish to reduce or stop alcohol consumption.
* Generally healthy with no unstable medical conditions, as determined by medical history, physical examination, routine blood labs, electrocardiogram, urine analysis, and urine toxicology.

Exclusion Criteria:

* Diagnosed with or having a family history of any of the following concomitant psychiatric disorders: schizophrenia or prodromal symptoms, any bipolar disorder, obsessive compulsive disorder, or other psychotic episode. Recent (within last 12 months) diagnosis of a major depressive disorder (MDD) (HAM-D score >19), treatment resistant depression (TRD), post-traumatic stress disorder (PTSD), panic disorder, or eating disorders.
* Subjects deemed unfit for psilocybin-assisted therapy based on the assessments made during psychotherapy sessions prior to the first psilocybin-assisted psychotherapy session.
* History of hallucinogen use disorder, or any use in the past 1 year, or >25 lifetime uses.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in the number of Heavy Drinking Days | 8 weeks
  Mean number of HDD from V5 (baseline) measured monthly (4 weeks) over the treatment period (Week 8), where heavy drinking is defined as the consumption of ≥60 g alcohol/day (if male) or ≥40 g alcohol/day (if female).

CONTACTS AND LOCATIONS:
Overall Officials: Hannu Alho, MD, Principal Investigator — Addiktum Oy
Locations (12):
- Canada (8):
  - Sabi Mind, Calgary, Alberta
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - Centre for Neurology Studies, Surrey, British Columbia
  - University of British Columbia, Department of Psychiatry, BRAIN Lab, Vancouver, British Columbia
  - Centricity Research, Halifax, Nova Scotia
  - MacAnxiety Research Centre, Hamilton, Ontario
  - Department of Psychiatry, Queen's University, Kingston, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
- Finland (4):
  - Research Center Oxidi Oy / Addiktum Oy, Helsinki
  - A-Klinikka, Kouvola
  - Mentacare Oy, Oulu
  - Addiktum Oy, Turku